CLINICAL TRIAL: NCT04942860
Title: The Evaluation of Vitiligous Lesions Repigmentation After Topical Administration of Methotrexate in Patients With Active Vitiligo
Acronym: EVRAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Rafal Czajkowski, Clinical Professor, Nicolaus Copernicus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WL107
Record Dates: First submitted 2021-06-02; First posted 2021-06-29 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Non-segmental Vitiligo
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Methotrexate 1% gel (Active Comparator): 1% methotrexate gel applied onto a predefined limb
  Interventions: Drug: 1% Methotrexate gel
- Methotrexate 0.5% gel (Active Comparator): 0.5% methotrexate gel applied onto a predefined limb
  Interventions: Drug: 0.5% Methotrexate gel
- Vehicle gel (Placebo Comparator): Vehicle gel applied onto a predefined limb
  Interventions: Drug: 1% Methotrexate gel; Drug: 0.5% Methotrexate gel

INTERVENTIONS:
Drug: 1% Methotrexate gel — 1% methotrexate gel applied onto a predefined limb
  Other Names: methotrexate
  Arms: Methotrexate 1% gel; Vehicle gel
Drug: 0.5% Methotrexate gel — 0.5% methotrexate gel applied onto a predefined limb
  Other Names: methotrexate
  Arms: Methotrexate 0.5% gel; Vehicle gel

SUMMARY:
The aim of this study is to evaluate the influence of two concentrations of methotrexate on vitiligous lesions in patients with non-segmental vitiligo

DETAILED DESCRIPTION:
Methotrexate, synthesized in the 1950s as an anticancer drug with an antiproliferative effect, is currently one of the most commonly used immunosuppressive agents in dermatology. The use of small, non-oncological doses has revealed its anti-inflammatory properties, including the impact on a number of cytokines involved in the pathogenesis of autoimmune diseases. It has been shown that treatment with methotrexate reduces the levels of TNF-alpha-producing T cells, while the number of IL-10 producing T cells increases. Methotrexate also inhibits the synthesis of interferon-γ. The above considerations justify the use of topical methotrexate in patients with vitiligo in order to obtain repigmentation.

A study has been designed as a single-center, randomized, double-blind, placebo-controlled pilot study with the enrollment of up to 100 active non-segmental vitiligo patients presenting with vitiligous lesions on both upper and lower limbs. Clinical effects of gel containing 1% methotrexate or 0.5% methotrexate applied on a preselected limb will be assessed in comparison with vehicle ointment applied on the opposite limb. All study participants will undergo clinical evaluation using Body Surface Area (BSA) and Vitiligo Area Scoring Index (VASI) scales at baseline, week 4, week 8 and week 12 time points. Precise assessment of skin lesions will be performed using photographic documentation obtained during each study visit and processed with NIS-Elements software.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of Clinic of Dermatology, Sexually Transmitted Diseases and Immunodermatology, Nicolaus Copernicus University, Collegium Medicum in Bydgoszcz
2. Provision of an informed consent form prior to any study procedures
3. Diagnosis of non-segmental acrofacial vitiligo with upper and lower limbs involvement
4. Active vitiligo, defined as appearance of new areas of depigmentation or progression of existing areas of depigmentation within 3 months preceding screening
5. Male or non-pregnant and non-breastfeeding female patients aged 18 to 80 years
6. Women must use effective contraception one month preceding treatment, during treatment and 6 months after completing treatment.
7. Confirmed valid health insurance

Exclusion Criteria:

1. Diagnosis of segmental, mixed, unclassified or undefined vitiligo
2. Pregnancy and breastfeeding
3. Hypersensitivity to methotrexate or any of the excipients
4. Systemic immunosuppressive/immunomodulating i.e. cyclosporine A, corticosteroids within 4 weeks preceding eligibility screening or azathioprine, methotrexate, mycophenolate mofetil, Janus kinase - JAK within 8 weeks preceding eligibility screening
5. Phototherapy due to vitiligo or any other medical conditions within the 4-week period preceding eligibility screening
6. Any topical or systemic additional vitiligo treatment (e.g. antioxidants, ginkgo biloba, dermo-cosmetics) within 4 weeks preceding screening
7. Surgical treatment of vitiligous lesions within past 4 weeks
8. Severe liver dysfunction [bilirubin> 5 mg / dL (85.5 μmol / L)], including cirrhosis and hepatitis
9. Severe renal impairment (eGFR <20 ml / min),
10. Disorders of the hematopoietic system, bone marrow disorders (leukopenia, thrombocytopenia, anemia),
11. Immunodeficiencies, including HIV infection
12. Severe acute or chronic infections such as tuberculosis
13. Alcohol abuse
14. Mouth ulcers and known active gastric or duodenal ulcer disease
15. Recent surgical wounds.
16. Skin malignancies (currently or history of skin malignancy within 5 years preceding screening)
17. Presence of skin characteristics that may interfere with study assessments
18. Patients currently participating in any other clinical study
19. Uncooperative patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
evaluation of repigmentation of vitiligous lesions achieved after the administration of 1% methotrexate or 0.5% methotrexate gels compared to vehicle gel after a 12-week study period | 12 weeks
  change from baseline in repigmentation on BSA scale at 12 weeks
evaluation of repigmentation of vitiligous lesions achieved after the administration of 1% methotrexate or 0.5% methotrexate gels compared to vehicle gel after a 12-week study period | 12 weeks
  change from baseline in repigmentation on VASI scale at 12 weeks

SECONDARY OUTCOMES:
percentage of patients who achieved particular response rate as follows none 0%; poor 1-25%; moderate 26-50%; good 51-75%; excellent >75% in each arm assessed as a relative reduction in BSA scale | 12 weeks
  number of: poor 1-25%; moderate 26-50%; good 51-75%; excellent >75% responders in each arm assessed as a relative reduction in BSA scale
percentage of patients who achieved particular response rate as follows none 0%; poor 1-25%; moderate 26-50%; good 51-75%; excellent >75% in each arm assessed as a relative reduction in VASI scale | 12 weeks
  number of: poor 1-25%; moderate 26-50%; good 51-75%; excellent >75% responders in each arm assessed as a relative reduction in VASI scale
comparison of 1% methotrexate and 0.5% methotrexate gel efficacy between study participants | 12 weeks
  comparison of BSA scale change between study arms
comparison of 1% methotrexate and 0.5% methotrexate gel efficacy between study participants | 12 weeks
  comparison of VASI scale change between study arms
the association between disease duration and repigmentation rate in study arms | 12 weeks
  the association between disease duration and repigmentation rate in study arms
rate of adverse events during treatment as assessed by CTCAE v4.0 | 12 weeks
  number of adverse events related to study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Czajkowski, Prof., Principal Investigator — Head of Chair and Clinic of Dermatology, Sexually Transmitted Diseases and Immunodermatology, Nicolaus Copernicus University in Torun, Ludwik Rydygier Medical College in Bydgoszcz
Locations (1):
- Clinic of Dermatology, Sexually Transmitted Diseases and Immunodermatology, Nicolaus Copernicus University, Faculty of Medicine in Bydgoszcz, Bydgoszcz, Cuiavian-Pomeranian, Poland

IPD SHARING:
Plan to Share IPD: No